CLINICAL TRIAL: NCT05683405
Title: Management of Peri-implantitis: Non-surgical Treatment of Peri-implantitis: Mechanical Debridement vs. Air-polishing
Brief Title: Management of Peri-implantitis: Non-surgical Treatment of Peri-implantitis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tannhelsetjenestens Kompetansesenter for Nord-Norge (Other)
Collaborators: Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 343997
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Peri-Implantitis
Keywords: Peri-implantitis; Non-surgical treatment; Air-polishing; Mechanical debridement; Bleeding on probing; periodontal pocket depth
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Each participant will be randomized to non-surgical treatment of peri-implantitits with either mechanical debridement or with air-polishing.
Who Masked: Outcomes Assessor
Masking Description: A periodontist that is not involved in the treatment and who is blinded to the treatment received will evaluate the treatment results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical debridement (Experimental)
  Interventions: Procedure: Non-surgical treatment of peri-implantitis with mechanical debridement
- Air polishing (Experimental)
  Interventions: Procedure: Non-surgical treatment of peri-implantitis with air polishing

INTERVENTIONS:
Procedure: Non-surgical treatment of peri-implantitis with mechanical debridement — Non-surgical treatment of peri-implantitis with mechanical debridement .
  Arms: Mechanical debridement
Procedure: Non-surgical treatment of peri-implantitis with air polishing — Non-surgical treatment of peri-implantitis with air polishing
  Arms: Air polishing

SUMMARY:
The goal of this clinical trial is to compare non-surgical treatment by mechanical debridement with air-polishing in peri-implantitis. The main question it aims to answer is:

• Does non-surgical treatment of peri-implantitis with an air-polishing devise (Perioflow® EMS, Nyon Switzerlad) provide a better treatment result than conventional cleaning with mechanical instruments?

Participants will receive non-surgical treatment of peri-implantitis either with mechanical debridement and with an air-polishing devise.

Researchers will compare pocket depth and bleeding/suppuration on probing in implants treated with the two methods to see if either of them is more efficient in treatment of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Referred to TkNN (Tannhelsetjenestens kompetansesenter for Nord-Norge) for treatment of peri-implantitis
* Participants should have at least one implants with peri-implantitis according to the diagnostic criteria from the 2017 Chicago Consensus Meeting.

Exclusion Criteria:

* Cemented prosthetic reconstructions, individuals smoking more than 10 cigarettes per day, individuals with diabetes and poor control of blood glucose levels, antibiotic treatment during the past threee months, and implants that are preferably to be extracted due to prognosis or function, are excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Probing depth | 26 weeks
  Probing depth 5 millimeters or more
Bleeding on probing | 26 weeks
  Bleeding from pocket on pocket depth probing
Suppuration on probing | 26 weeks
  Suppuration from pocket on pocket depth probing

CONTACTS AND LOCATIONS:
Locations (1):
- Tannhelsetjenestens kompetansesenter for Nord-Norge, Tromsø, Troms, Norway